CLINICAL TRIAL: NCT00553891
Title: Double Blind, Placebo Controlled Trial, Evaluating the Role of Nasonex® in the Management of Nasal Obstruction Secondary to Adenoids Hypertrophy in Children
Brief Title: Placebo-controlled Trial With Nasonex for Nasal Obstruction Secondary to Adenoids Hypertrophy in Children (P04367)(TERMINATED)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment because of war in the study country.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04367
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Nasal Obstruction; Adenoids Hypertrophy; Adenoidectomy
MeSH Terms: conditions — Nasal Obstruction | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasonex Nasal Spray (Experimental)
  Interventions: Drug: mometasone furoate nasal spray
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Drug: placebo nasal spray

INTERVENTIONS:
Drug: mometasone furoate nasal spray — One spray (50 mcg per spray) in each nostril once daily (100 mcg daily) for 3 months.
  Other Names: SCH 32088; Nasonex
  Arms: Nasonex Nasal Spray
Drug: placebo nasal spray — One spray in each nostril once daily for 3 months.
  Arms: Placebo Nasal Spray

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to document the long-term effect of treatment with mometasone furoate nasal spray in moderate to severe adenoids hypertrophy as reflected by the need for removal of the adenoids within one year of the treatment regimen. Subjects will be assigned treated with either mometasone furoate nasal spray or placebo for 3 months. Subjects will be followed for an addition 12 months. Serious AEs will be followed starting first dose-till 30 days after study treatment period completion.

This study was terminated - Please see "P04367 - Lebanon"

ELIGIBILITY:
Inclusion Criteria:

* Should be between 2 and 11 years.
* Should have nasal obstruction for at least 3 months.
* Should have evidence of adenoids hypertrophy by nasopharyngoscopy, which cause >50% obstruction of the posterior choanae.
* May have concomitant allergic rhinitis, by history, & and specific blood studies; however, the symptoms should be under control during the study period.

Exclusion Criteria:

* Patients with less than 50% obstruction of the post choanae.
* Patients with history of recurrent epistaxis or immunodeficiency.
* Patients with severe septal deviation.
* Patients with unilateral or bilateral choanal atresia, large nasal polyps or any nasal mass.
* Known allergy to the drug.
* Presence of chronic otitis media defined as: otorreha + perforation (concomitant otitis media with effusion, or recurrent otitis media are not excluded).
* Cystic fibrosis & other causes responsible for nasal obstruction.
* Infection (ie; sinusitis).
* History of recent surgery or trauma to nose, unless all wounds have healed.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To document the long-term effect of treatment with Nasonex in moderate to severe adenoids hypertrophy (which cause >50% obstruction of the posterior choanae). as reflected by the need for adenoidectomy within one year of the treatment regimen. | The total duration of therapy is 3 months the follow up period is for 12 months.

SECONDARY OUTCOMES:
To identify the characteristics of subjects who will show complete or significant resolution of the nasal obstruction symptoms secondary to enlarged adenoids, upon using Nasonex. | The total duration of therapy is 3 months the follow up period is for 12 months.